CLINICAL TRIAL: NCT00119093
Title: Home-based AIDS Care Project, Tororo, Uganda
Brief Title: Home-based AIDS Care Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by IRB for non-compliance with human subject regulations.
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: The AIDS Support Organization (Other); Ministry of Health, Uganda (Other Government)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-3666
Record Dates: First submitted 2005-07-08; First posted 2005-07-13 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: Antiretroviral therapy; HIV; Adherence; Viral Load; Opportunistic illness
MeSH Terms: conditions — HIV Infections | interventions — Laboratories

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Laboratory and clinical monitoring regimens

SUMMARY:
The Home-based AIDS care program pilot project delivers and monitors antiretroviral (ARV) and tuberculosis (TB) medications at the homes of 1,000 people with HIV living in a rural area of Uganda. This study is evaluating how well this program reduces illness and prolongs the life of participants, changes sexual behavior, influences levels of adherence to medication, affects aspects of perceived stigma by participants and their communities, and other operational components of the program including cost-effectiveness. This study is evaluating the hypothesis that frequent home visits by a trained lay person with a standard questionnaire is equivalent in terms of health outcomes to frequent viral load and CD4 cell count measurements.

DETAILED DESCRIPTION:
In Uganda, the high cost and complexity of administering antiretroviral therapy is an obstacle to full implementation country-wide. The Home-based AIDS care program (HBAC) pilot project was designed to deliver and monitor ARV and tuberculosis (TB) medications at the homes of 1,000 people with HIV living in a rural area of Uganda. In addition, the cost and complexity of frequent laboratory monitoring of viral load and CD4 cell counts is a major impediment to widespread use of ARV therapies in Uganda and other resource-limited settings. Nested within the Home-Based AIDS Care (HBAC) project, is a randomized study of strategies for monitoring ARV therapy that involves 3 arms: 1) Quarterly CD4 cell counts, viral loads and home visits by trained lay persons; 2) Quarterly CD4 cell counts and home visits; and 3) Home visits alone.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* CD4 cell count <250 or symptomatic AIDS
* Age >13 years
* Karnofsky score >40%
* AST or ALT < 5 times normal values
* Creatinine clearance >25 ml/min

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2003-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Equivalence of 3 different monitoring regimens for ART

SECONDARY OUTCOMES:
Sexual risk behavior
medication adherence
quality of life
depression
cost-effectiveness
viral load
CD4 cell count

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Bunnell, ScD, MEd, Principal Investigator — Centers for Disease Control and Prevention; Jonathan H Mermin, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Alex Coutinho, MBChB, MPH, Principal Investigator — The AIDS Support Organization; David Moore, MD, Principal Investigator — CDC-Uganda and University of British Columbia; Jordan Tappero, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Tororo Hospital/CDC-Uganda, Tororo, Tororo, Uganda

REFERENCES:
- [Derived] Ekwaru JP, Campbell J, Malamba S, Moore DM, Were W, Mermin J. The effect of opportunistic illness on HIV RNA viral load and CD4+ T cell count among HIV-positive adults taking antiretroviral therapy. J Int AIDS Soc. 2013 Apr 1;16(1):17355. doi: 10.7448/IAS.16.1.17355. PMID 23547778
- [Derived] Campbell JD, Moore D, Degerman R, Kaharuza F, Were W, Muramuzi E, Odongo G, Wetaka M, Mermin J, Tappero JW. HIV-infected ugandan adults taking antiretroviral therapy with CD4 counts >200 cells/muL who discontinue cotrimoxazole prophylaxis have increased risk of malaria and diarrhea. Clin Infect Dis. 2012 Apr;54(8):1204-11. doi: 10.1093/cid/cis013. Epub 2012 Mar 14. PMID 22423133
- [Derived] Mermin J, Ekwaru JP, Were W, Degerman R, Bunnell R, Kaharuza F, Downing R, Coutinho A, Solberg P, Alexander LN, Tappero J, Campbell J, Moore DM. Utility of routine viral load, CD4 cell count, and clinical monitoring among adults with HIV receiving antiretroviral therapy in Uganda: randomised trial. BMJ. 2011 Nov 9;343:d6792. doi: 10.1136/bmj.d6792. PMID 22074711
- [Derived] Weidle PJ, Moore D, Mermin J, Buchacz K, Were W, Downing R, Kigozi A, Ndazima V, Peters P, Brooks JT. Liver enzymes improve over twenty-four months of first-line non-nucleoside reverse transcriptase inhibitor-based therapy in rural Uganda. AIDS Patient Care STDS. 2008 Oct;22(10):787-95. doi: 10.1089/apc.2008.0020. PMID 18778241